CLINICAL TRIAL: NCT01727570
Title: Prehabilitation to Overcome the Stress of Surgery: the Role of Nutrition in Enhancing Postoperative Functional Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franco Carli (Other)
Collaborators: Immunotec Inc. (Industry)
Responsible Party: Sponsor-Investigator, Franco Carli, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 11-240-SDR
Record Dates: First submitted 2012-10-31; First posted 2012-11-16 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Colorectal Cancer
Keywords: Cancer; Colon; Rectum; Surgery
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrition Counselling (No Intervention): Patients will be asked to fill out a three day record of all food and drink consumed. Patients will be given an appointment with the nutritionist approximately 4 weeks before surgery to go over their regular diet and advice will be given on how to improve the nutritional quality of their diet
- Nutrition Supplementation (Active Comparator): Patients will be asked to fill out a three day record of all food and drink consumed. An appointment with the nutritionist will be given approximately 4 weeks before surgery to go over their regular diet and advice will be given on how to improve the nutritional quality of the diet. Patients will also be given a supply of nutritional supplements to take orally (by mouth) every day. These supplements include a whey protein isolate (Immunocal®, Immunotec Inc), omega-3 fatty acids from fish oil, and vitamins/minerals.
  Interventions: Dietary Supplement: Whey Protein (Immunocal®)

INTERVENTIONS:
Dietary Supplement: Whey Protein (Immunocal®) — The amount of Immunocal® whey protein the patient is required to take daily will be determined on an individual basis by the nutritionist according to the assessed protein deficit in the patient's diet.
  Arms: Nutrition Supplementation

SUMMARY:
To determine the impact of nutritional supplementation with whey protein on postoperative functional capacity in patients undergoing colorectal surgery for cancer.It is hypothesized that, compared with a control group receiving nutrition counselling only, patients receiving nutritional counselling along with preoperative and postoperative nutritional supplements will have a significantly improved change in functional walking capacity from baseline to 8 weeks after surgery.

DETAILED DESCRIPTION:
The aims of this research project are the following:

1. Determine to what extent a nutritional prehabilitation regimen, which includes whey protein, initiated before surgery and continued after surgery, optimizes the recovery of functional walking capacity following colorectal resection for cancer.
2. To understand further which measures of immediate surgical recovery are sensitive to prehabilitation interventions, and predict change in later outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* +18 years of age
* referred electively for resection of malignant, non metastasized, colorectal lesions
* French or English speaking

Exclusion Criteria:

* ASA class 4-5
* co-morbid medical, physical and mental conditions (e.g.dementia, disabling orthopedic and neuromuscular disease, psychosis)
* cardiac abnormalities
* severe end-organ disease such as cardiac failure (New York Heart Association classes I-IV), COPD, renal failure (creatinine > 1.5 mg/dl, and hepatic failure ALT and AST >50% over the normal range)
* sepsis
* morbid obesity (BMI >40)
* anemia (hematocrit < 30 %, haemoglobin <10g/dl, albumin < 25mg/dl).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Six-Minute Walk Test (6MWT) | up to 8 weeks after surgery
  Change in functional walking capacity will be assessed throughout the study according to the 6-Minute Walk Test (6MWT). The 6MWT evaluates the ability of an individual to maintain a moderate level of physical activity over a time period reflective of the activities of daily living. Subjects are instructed to walk back and forth, in a 20 m stretch of hallway, for six minutes, at a pace that would make them tired by the end of the walk; encouragement and feedback are given according to published guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Gillis C, Nguyen TH, Liberman AS, Carli F. Nutrition adequacy in enhanced recovery after surgery: a single academic center experience. Nutr Clin Pract. 2015 Jun;30(3):414-9. doi: 10.1177/0884533614562840. Epub 2014 Dec 29. PMID 25547338